CLINICAL TRIAL: NCT06916325
Title: DeLIVER Trial: A Prospective, Multi-Center, Single-Arm, Open Label Trial of Deceased Donor Livers Transplanted After DHOPE With eXVIVO LIVER Perfusion
Brief Title: Open Label Trial of Deceased Donor Livers Transplanted After DHOPE With eXVIVO LIVER Perfusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: XVIVO Perfusion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LiA-US-001
Record Dates: First submitted 2025-03-21; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Liver Transplant Surgery; Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Participants requiring liver transplant (Experimental): Extended criteria donor donation after brain death (ECD-DBD) or donation after circulatory death (DCD) donor organs will be recovered, transported via static cold storage (SCS), and undergo dual hypothermic oxygenated perfusion (DHOPE) on Liver Assist.
  Interventions: Device: dual hypothermic oxygenated perfusion (DHOPE)

INTERVENTIONS:
Device: dual hypothermic oxygenated perfusion (DHOPE) — Clinically, end-ischemic DHOPE has been shown to restore hepatic ATP, reduce reperfusion injury, and improve outcomes after deceased donor liver transplantation. Recent prospective and retrospective clinical studies detail the safety and feasibility of prolonged preservation of donor livers with DHOPE for up to 20 hours; prolonged perfusion has shown similarly low rates of serious adverse events, a potential protective effect in mitigating acute kidney injury and may facilitate decreased frequency of discarded and nonuse of donor livers.

SUMMARY:
The purpose of this clinical study is to confirm the safety and effectiveness of dual hypothermic oxygenated perfusion (DHOPE) using the Liver Assist to preserve deceased donor livers for transplantation.

ELIGIBILITY:
Participant Inclusion Criteria:

1. Participant is able to provide informed consent and HIPAA authorization
2. Age ≥18 years
3. Participant is registered as an active first-time liver transplant candidate on the United Network for Organ Sharing (UNOS) waiting list for primary liver transplantation

   - For participants with hepatocellular carcinoma (HCC) as indication for Orthotopic Liver Transplantation, the tumor must be within Milan Criteria or down-staged to Milan Criteria at the time of transplant
4. Participant is willing to comply with the study requirements and procedures

Participant Exclusion Criteria:

1. Participant will undergo concurrent multi-organ transplantations (liver-kidney, liver-lung, etc.)
2. Participant is listed for liver transplantation due to fulminant liver failure (UNOS status 1A)
3. Participant is listed for a repeat liver transplantation (>1 graft)
4. Participant is pregnant
5. Participant is on respiratory (ventilator dependent) and/or cardiocirculatory support (defined as mechanical circulatory support which requires at least one intravenous inotrope to maintain hemodynamics)
6. Participant is enrolled in an interventional clinical trial with an investigational drug or device
7. Presence of other medical, social, or psychological conditions that in the investigator's opinion, could limit the participant's ability to participate in the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Early Allograft Dysfunction | Day 7 (post operative)
  Incidence of Early Allograft Dysfunction (EAD) defined according to the Olthoff criteria as the presence of one or more of the following postoperative laboratory analyses observations reflective of liver injury and function:
  * Bilirubin ≥ 10mg/dL on postoperative day (POD) 7, or
  * International normalized ratio (INR) ≥ 1.6 on POD 7, or
  * Alanine or aspartate aminotransferases (AST and ALT) > 2000 IU/L within the first 7 PODs
Overall graft survival | Day 180 (post operative)
  Overall graft survival

IPD SHARING:
Plan to Share IPD: No